CLINICAL TRIAL: NCT03217032
Title: Lentiviral FVIII Gene Therapy for Hemophilia A
Brief Title: Lentiviral FVIII Gene Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17007
Record Dates: First submitted 2017-07-03; First posted 2017-07-13 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; factor VIII; Gene therapy; lentiviral vector
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YUVA-GT-F801 (Experimental): Gene transfer to treat Hemophilia A
  Interventions: Biological: YUVA-GT-F801

INTERVENTIONS:
Biological: YUVA-GT-F801 — Lentiviral factor VIII gene modified autologous hematopoeitic stem cells and mesenchymal stem cells

SUMMARY:
This study is a Phase I trial using an advanced lentiviral vector to deliver a functional gene for human clotting factor VIII into patients with hemophilia A, to evaluate the safety and efficacy of infusion of lentiviral gene modified autologous stem cells in patients.

DETAILED DESCRIPTION:
Hemophilia A is a genetic bleeding disorder caused by the lack of ability to produce blood-clotting factor VIII (FVIII). Individuals with hemophilia A suffer repeated bleeding episodes, which can cause chronic joint disease and sometimes even death due to the inability for blood to clot efficiently. The current treatment is intravenous infusion of clotting factor concentrates, either prophylactically or in response to bleeding. The procedure is life time long and expensive while still cannot achieve a cure.Gene therapy is a novel technology that has been successfully demonstrated in a number of clinical studies for diseases such as cancer and genetic diseases. In this study, an advanced lentiviral vector system NHP/TYF will be used to deliver a functional FVIII gene to overcome human clotting FVIII gene defect in patients with hemophilia A. This study is a Phase I trial evaluating the safety and efficacy for infusion of gene modified autologous stem cells in patients with hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent and comply with requirements of the study.
2. Males ≥2 years with confirmed diagnosis of hemophilia A (endogenous factor VIII ≤2 IU/dL or ≤2% of normal).
3. A minimum average of 4 bleeding events per year requiring episodic treatment of factor VIII infusions or prophylactic factor VIII infusions.
4. No measurable factor VIII inhibitor as assessed by the central laboratory and have no prior history of inhibitors to factor VIII protein.
5. Agree to use reliable barrier contraception until 3 consecutive samples are negative for vector sequences.

Exclusion Criteria:

1. Significant liver dysfunction as defined by abnormal alanine transaminase, bilirubin and alkaline phosphatase.
2. History of inhibitor against factor VIII.
3. Evidence of active hepatitis B or C and currently on antiviral therapy.
4. Have serological evidence of HIV-1 or HIV-2 with CD4 counts ≤200/mm3 (subjects who are HIV+ and stable with CD4 count >200/mm3 and undetectable viral load are eligible to enroll).
5. Any evidence of active infection or any immunosuppressive disorder.
6. Participated in a gene transfer trial within the last 6 months or in a clinical trial with an investigational drug within the last 12 weeks.
7. Unable or unwilling to comply with study assessments.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing drug-related adverse events | a year
  As assessed by physical exam, vital signs, standard clinical labs, and Bethesda assay for FVIII inhibitor

SECONDARY OUTCOMES:
Changes from baseline in circulating FVIII activity (IU/dL or % normal) | a year

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No